CLINICAL TRIAL: NCT06251700
Title: Longterm Effectiveness of Artificial Intelligence-assisted Colonoscopy on Adenoma Recurrence - a Prospective Longitudinal Follow-up of Randomized Controlled Trial
Brief Title: Longterm Effectiveness of Artificial Intelligence-assisted Colonoscopy on Adenoma Recurrence
Acronym: ENDOAID-PRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023.541
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Screening Colonscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental): CADe system will be used during withdrawal phase of colonscopy
  Interventions: Device: ENDO-AID CADe

INTERVENTIONS:
Device: ENDO-AID CADe — ENDO-AID CADe will be used during the withdrawal process of the colonscopy

SUMMARY:
We hypothesize that AI-assisted colonoscopy can reduce post-colonoscopy neoplasia incidence after 3 years, over standard colonoscopy. Moreover, this protective effect may allow surveillance intervals to be lengthened, by modifying long-term outcome of high-risk subgroup.

DETAILED DESCRIPTION:
Between April 2021 and July 2022, our group completed a parallel-group, randomized controlled trial in Hong Kong. [ENDOAID-TRAIN study; NCT04838951] 856 subjects undergoing colonoscopies were randomized 1:1 to receive colonoscopies with CADe (ENDO-AID, Olympus Co., Japan) or standard colonoscopies (control). Our study proved that AI-assisted colonoscopies could increase the overall ADR, especially small-to-medium size adenomas. It remains questionable whether the increased detection and removal of these non-advanced adenomas can be translated into any sustained long-term benefit. The impact of this AI-driven intensive surveillance on general population and healthcare system is also largely unknown. In this research project, we aim to assess the long-term effectiveness of AI-assisted colonoscopy on adenoma recurrence and PCCRC prevention, by conducting a real-world, prospective study with longitudinal extension from a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible if:

(i) They underwent randomization to receive colonoscopy with/without CADe in ENDOAID-TRAIN study [NCT04838951]; (ii) They are fit and willing to undergo surveillance colonoscopy at year 3; (iii) Written informed consent obtained.

Exclusion Criteria:

Subjects will be excluded from the study if they have any of the followings:

(i) Incomplete colonoscopy during index procedure; (ii) Known residual colorectal neoplasia not removed (except hyperplastic polyps); (iii) Underwent unscheduled interval colonoscopy before year 3; (iv) Contraindications to surveillance colonoscopy at year 3; (v) Advanced comorbid (American Society of Anesthesiologists grade 4 or above); (vi) History of CRC, hereditary polyposis syndrome or inflammatory bowel disease; (vii) History of colectomy at any time point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 775 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Post-colonoscopy adenomas at year 3 | During the colonoscopy
  The primary endpoint is the incidence of post-colonoscopy adenomas at year 3, which is the composite of new occurrence and metachronous recurrence of adenomas during surveillance.

SECONDARY OUTCOMES:
Post-colonoscopy AA | During the colonoscopy
  Incidence of post-colonoscopy advanced adenomas
Post-colonoscopy advanced neoplasms | During the colonoscopy
  Incidence of post-colonoscopy advanced neoplasms
Post-colonoscopy SSL | During the colonoscopy
  Incidence of post-colonoscopy SSL
Post-colonoscopy CRC | During the colonoscopy
  Incidence of post-colonoscopy CRC
Post-colonoscopy adenomas and advanced adenomas | During the colonoscopy
  Number of post-colonoscopy adenomas and advanced adenomas
Size and location of post-colonoscopy adenomas and advanced adenomas | During the colonoscopy
  Size and location of post-colonoscopy adenomas and advanced adenomas
High-risk and low-risk group according to USMSTF guideline | During the colonoscopy
  Proportion of subjects re-classified as high-risk and low-risk groups according to USMSTF guideline

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No